CLINICAL TRIAL: NCT01881269
Title: Assessment of Respiration Rate Monitoring During Transitions From Spontaneous to Controlled Ventilation
Brief Title: Respiration Rate Monitoring During Transitions
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0409
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Focus of the Study is Measuring Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: No treatment, prospective observational

SUMMARY:
The purpose of this study is to evaluate the performance of the software that calculates respiration rate for the study pulse oximetry monitoring system during transitions of ventilation type from spontaneous breathing to controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Be undergoing a procedure with planned general anesthesia involving placement of an endotracheal tube or laryngeal mask airway following induction of anesthesia.
* American Society of Anesthesiologists physical status classification (ASA) Status 1, 2 or 3.
* Body mass index (BMI) ≤30 kg/m2.
* Subject is willing and able to provide written consent.

Exclusion Criteria:

* Female subjects of child-bearing potential with a positive pregnancy test or an absence of documented non-childbearing status in the medical history records.
* Female subjects who are currently lactating and breastfeeding.
* Subjects with any evidence of potential difficulty in mask ventilation and/or tracheal intubation.
* Subject has an abnormality that may prevent proper application of the device/sensors.
* Subject is in atrial fibrillation.
* Subject has a documented history of frequent premature ventricular contractions (PVCs), defined as greater than 3 in 30 seconds or greater than 6 in 60 seconds.
* Subject has an implanted pacemaker.
* Subjects with non-sinus rhythm, frequent premature ventricular complexes (> 5 min), or abnormal PR, QRS, or QT intervals on screening ECG.
* Subjects with artificial finger nails.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects from a hospital population, who are scheduled to undergo surgery requiring general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Time to report a Respiration Rate value after initiation of controlled ventilation | 1 - 3 minutes after the initiation of controlled ventilation
  Time (in seconds) for the software to report a Respiration Rate value within one breath per minute of the controlled ventilation rate after placement of the airway device (endotracheal tube or laryngeal mask airway)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lumbley, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States